CLINICAL TRIAL: NCT02892539
Title: A Prospective Multicenter Case Study to Evaluate Radiation Exposure and Risk Factors in Patients During Coronary Angiography
Brief Title: Evaluation of Radiation Exposure and Risk Factors During Coronary Angiography
Acronym: EARTH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fan Liu (Other)
Collaborators: The First Hospital of Hebei Medical University (Other); Hebei Medical University Third Hospital (Other); Hebei Medical University Fourth Hospital (Other); Bethune International Peace Hospital (Other); First Hospital of Shijiazhuang City (Other); Xingtai People's Hospital (Other); Cangzhou Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Fan Liu, Director of Department of Cardiology, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Other Study IDs: Hebei Tracking Project 2016
Record Dates: First submitted 2016-08-27; First posted 2016-09-08 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Coronary Angiography

SUMMARY:
The purpose of this study is to evaluate the radiation exposure in patients undergoing coronary angiography, and to identify reference values for the main radiation doses parameters.

DETAILED DESCRIPTION:
Exposure of patients to X-rays during interventional coronary procedures may have deleterious effects, including an increased risk of developing cancer.Individual justification for the procedure and its optimization are the cornerstones of dose-reduction for patients.Radiation exposure is influenced by a variety of technical and clinical factors.Few multicenter data from large populations exist concerning the radiation doses to which patients are exposed during interventional coronary procedures.The aims of this prospective, multicenter survey is to: 1) evaluate the radiation exposure in 4000 patients undergoing coronary angiography by monitoring the parameters of Air kema,fluoroscopy Dose-area product and total Dose-area product; 2) analyze factors associated with variation in radiation dose in everyday clinical practice, such as number of frames, body surface area, sex, age, BMI, arterial approach, fluoroscopy time and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need to perform coronary angiography

Exclusion Criteria:

* Contrast medium reactions Severe cardiopulmonary insufficiency Uncontrolled severe arrhythmia Uncorrected kaliopenic, digitalism and acid-base imbalance Severe liver and renal dysfunction Hemorrhagic disease Severe infection disease Others who were unwilling to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: residents who need to perform coronary angiography in Hebei province
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure of the patients | during coronary angiography procedure

SECONDARY OUTCOMES:
Reference values for the main radiation doses parameters | during coronary angiography procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fan Liu, MD/PhD, Principal Investigator — The Second Hospital of Hebei Medical Univerisity
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Result] Shah A, Das P, Subkovas E, Buch AN, Rees M, Bellamy C. Radiation dose during coronary angiogram: relation to body mass index. Heart Lung Circ. 2015 Jan;24(1):21-5. doi: 10.1016/j.hlc.2014.05.018. Epub 2014 Jun 23. PMID 25065542
- [Result] Wassef AW, Hiebert B, Ravandi A, Ducas J, Minhas K, Vo M, Kass M, Parmar G, Hussain F. Radiation dose reduction in the cardiac catheterization laboratory utilizing a novel protocol. JACC Cardiovasc Interv. 2014 May;7(5):550-7. doi: 10.1016/j.jcin.2013.11.022. Epub 2014 Apr 16. PMID 24746655